CLINICAL TRIAL: NCT01920009
Title: Feasibility and Potential Impact of Community Pharmacy Care Including Motivational Interviews on Adherence to Secondary Prevention Medication in Patients With Coronary Heart Diseases
Brief Title: Impact of Motivational Interviews Within Pharmacy Care Upon Adherence to Cardiovascular Medicines
Acronym: Pharmacycare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13/0064
Record Dates: First submitted 2013-08-05; First posted 2013-08-09 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Heart Disease
Keywords: pharmacy care; adherence; coronary heart disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacy care group (Active Comparator): patients in this group will receive two counseling sessions with a motivational interview.
  Interventions: Behavioral: Pharmacist counselling session with a motivational interview
- Controlgroup (No Intervention): patients in this group will receive usual care by pharmacists

INTERVENTIONS:
Behavioral: Pharmacist counselling session with a motivational interview — The intervention:
  The patient will be invited by the community pharmacist for two consultations the first 2 weeks after discharge and the second after 3 months.
  The intervention group consultation:
  Community pharmacy consultation around 2 weeks The consultation will take place in the pharmacy a face to face consultation for 20 minutes including; Motivational interview session, the pharmacists will incorporate the key motivational interview skills in their consultation "Express empathy, develop discrepancy, role with resistance, support self efficacy".
  The sessions will aim to develop a partnership between the pharmacist with the patient and exchange information to facilitate an informed decision. Furthermore both the pharmacist and the patient will negotiate behaviour and reach an agreement. The goal is to access motivation and elicit commitment to change behaviour "in this case would be adherence to life saving medication"
  Other Names: Two counseling sessions including a motivational interview; Medication usage review session including a motivational interview; New medicine service session including a motivational interview
  Arms: Pharmacy care group

SUMMARY:
Introduction:

In the United Kingdom(UK), about 838,000 men and 394,000 women have had a myocardial infarction (MI) and will need secondary prevention medications. Longterm adherence to secondary prevention therapies remains poor, nonadherence to medication in MI patients ranges from 13-60%(1). Studies show that approximately one fourth of cardiac patients do not refill their cardiac medications (2). Strategies to tackle the burden of non adherence could involve pharmacy care and The New Medicine Service (which is a service provided by community pharmacists to help patients on long term medications for chronic diseases) with a motivational interview incorporated as part of the counselling session of a community pharmacist. Communication of health providers with patients and between health providers could also be an important strategy to improve adherence.

Cardiovascular disease is high in all ethnic groups as well as in the general population; however it is the South Asians who have the highest prevalence of coronary heart disease (CHD) (3). In addition, South Asians develop CHD at a younger age, often before the age of 40 years (3).

Aim of this study:

This study is to investigate the feasibility and potential impact of a pharmacy care intervention involving motivational interviews and referral to the New Medicine Service in coronary heart disease patients on adherence to secondary prevention medication and on outcomes of coronary heart disease.

Method:

The study is designed as a prospective, controlled feasibility/pilot, intervention study. The study has two phases.

In the intervention phase a total of 200 coronary heart disease patients discharged from the London Chest Hospital will be enrolled into the study and followed up for one year. Pharmacies from up to six London Boroughs will be invited to take place in the study. Pharmacies will be randomised using a table of random numbers into intervention site or control site. The pharmacists working in the intervention pharmacies will be invited for training on the delivery of the intervention and on motivational interviewing. The intervention will be performed by community pharmacists. Recruitment of patients will take place in the hospital. In the interview phase 20 patients from South Asian backgrounds will be invited for a telephone interview to study the effect of their beliefs and cultural backgrounds in regards to their adherence to cardiac medication.

Outcome measures:

The primary outcome measure is self report adherence with coronary artery disease medication employing a standard validated measure. Secondary outcomes are blood pressure and LDL-C (low density lipoprotein cholesterol) in addition to data regarding the feasibility of the intervention.

Analysis:

Both quantitative and qualitative data analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18-yr-old.
* Both Male/female.
* Acute coronary syndromes; angina, NSTEMI (non-ST-segment elevation myocardial infarction) /unstable angina, STEMI (ST segment elevation myocardial infarction).
* Patients included are from high risk group (hypertension , diabetes, hyperlipidemia), as well as patient from low risk group (developed MI with an unknown risk factor).
* Patients medically treated for secondary prevention of coronary artery disease (dual antiplatelet therapy aspirin plus either clopidogrel, ticagrelor or prasugrel. Beta-blockers, or calcium channel blockers, ACE-inhibitors or ARBs (angiotensin II receptor blocker), and statins).
* Patients living in the area around East London and who regularly refill prescriptions in the pharmacies involved in the study.

Exclusion Criteria:

* Congenital heart disease.
* Complications of myocardial infarction: Arrhythmias, Congestive Heart Failure, Tamponade / Thromboembolic disorder, Rupture (Ventricle, septum, papillary muscle), Aneurysm (Ventricle), Pericarditis, Infection.
* Patients who do not live in the area around East London and do not regularly refill prescriptions in the pharmacies involved in the study.
* Patients who do not live independently (living or nursing home residence).
* Patients with less than one year survival rate.
* Patients unable to understand oral and written English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in adherence to cardiovascular medication | Change in adherence from baseline assessed at 6 months and 12 months.

SECONDARY OUTCOMES:
Change in blood pressure and LDL-C. | Change in blood pressure and LDL-C from baseline assessed at 6 months and 12 months.
Cost of the intervention. | 6 months
  Cost of the intervention: This will include training of the community pharmacists on motivational interviews. Cost of the community pharmacist intervention in terms of time and material spent on counselling patients and establish if this can be accommodated into a daily schedule of a community pharmacy and how many sessions can one pharmacy manage per day.

OTHER OUTCOMES:
Patient satisfaction/feedback on the pharmacist intervention | 6 months
  This will be assessed by semi-structured telephone interviews conducted by the research pharmacist.

CONTACTS AND LOCATIONS:
Overall Officials: Felicity Smith, Professor, Study Director — UCL-School of Pharmacy; David Taylor, Professor, Study Chair — UCL-School of Pharmacy; Consultant Pharmacist Sotiris Antoniou, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- The London Chest Hospital, London, London, United Kingdom

REFERENCES:
- [Background] Garavalia L, Garavalia B, Spertus JA, Decker C. Exploring patients' reasons for discontinuance of heart medications. J Cardiovasc Nurs. 2009 Sep-Oct;24(5):371-9. doi: 10.1097/JCN.0b013e3181ae7b2a. PMID 19707097
- [Background] Jackevicius CA, Li P, Tu JV. Prevalence, predictors, and outcomes of primary nonadherence after acute myocardial infarction. Circulation. 2008 Feb 26;117(8):1028-36. doi: 10.1161/CIRCULATIONAHA.107.706820. PMID 18299512
- [Background] Gupta M, Singh N, Verma S. South Asians and cardiovascular risk: what clinicians should know. Circulation. 2006 Jun 27;113(25):e924-9. doi: 10.1161/CIRCULATIONAHA.105.583815. No abstract available. PMID 16801466
- [Derived] M A Jalal ZS, Smith F, Taylor D, Finlay K, Patel H, Antoniou S. Impact of pharmacy care upon adherence to cardiovascular medicines: a feasibility pilot controlled trial. Eur J Hosp Pharm. 2016 Sep;23(5):250-256. doi: 10.1136/ejhpharm-2015-000790. Epub 2016 Feb 2. PMID 31156861